CLINICAL TRIAL: NCT04224181
Title: Inflammation and Cardiovascular Health in Women
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Markella V. Zanni,M.D., Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2019P001220
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: HIV/AIDS; Myocardial Infarction
Keywords: Women; Arterial Inflammation; Systemic Immune Activation; Endothelial Dysfunction; Cardiovascular Disease Risk
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Myocardial Infarction; Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, PBMCs, plasma, serum, endothelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with HIV: Individuals with female nascent sex who have been diagnosed with HIV.
  Interventions: Radiation: Cardiac PET; Radiation: 99mTc-tilmanocept SPECT/CT; Radiation: Contrast Enhanced Coronary and Aortic Computed Tomography Angiography
- Women without HIV: Individuals with female nascent sex who do not have HIV.
  Interventions: Radiation: Cardiac PET; Radiation: 99mTc-tilmanocept SPECT/CT; Radiation: Contrast Enhanced Coronary and Aortic Computed Tomography Angiography

INTERVENTIONS:
Radiation: Cardiac PET — A scan examining blood flow to the heart
Radiation: 99mTc-tilmanocept SPECT/CT — A scan to look at inflammation in the arteries
Radiation: Contrast Enhanced Coronary and Aortic Computed Tomography Angiography — A scan of the heart and surrounding blood vessels

SUMMARY:
Systemic immune activation and inflammation are believed to play a significant role in the development and clinical course of myocardial infarction (MI). Among women with HIV (WHIV), heightened systemic immune activation and inflammation persist, even when HIV infection is well-treated with contemporary antiretroviral therapeutic regimens. Moreover, WHIV in high-resource regions face a three-fold increased risk of myocardial infarction as compared with matched non-HIV-infected women. The goals of this study are to better understand ways in which HIV infection-incited systemic immune activation and inflammation augment MI risk among women.

DETAILED DESCRIPTION:
The goals of this study are to better understand ways in which HIV infection-incited systemic immune activation and inflammation augment MI risk among women. To this end, WHIV and non-HIV-infected women will undergo structural and functional cardiovascular imaging studies (Cardiac PET, 99mTc-tilmanocept SPECT/CT, Contrast Enhanced Coronary and Aortic Computed Tomography Angiography) as well as vascular, metabolic/hormonal, and immune phenotyping. Measures of immune activation, arterial inflammation, and cardiovascular pathology will be compared between groups and interrelationships between these parameters will be assessed among WHIV.

ELIGIBILITY:
WHIV:

Inclusion

* female nascent sex
* HIV
* age 40-79
* self-report of stable ART for at least 180 days prior to study entry - any regimen (no more than 30 days missed medication in the last 180 days)

Exclusion

* self-reported history of MI, stroke, coronary revascularization
* stable or unstable angina symptoms
* a pre-existing diagnosis of diabetes, being actively treated with oral or injectable antihyperglycemic medication
* current cocaine use
* current use of exogenous oral, or transdermal, injected, or depot estrogen or testosterone
* current treatment with prescription, systemic (oral, IV, or IM) steroids, or anti-inflammatory/immune suppressant medical therapies (excluding topical therapies, UV therapy, ASA-derivative therapies, or NSAIDs) for autoimmune/inflammatory diseases (psoriasis, RA, IBD, lupus), post-transplant care, asthma, or pain syndromes
* use of oral steroids or prescription oral anti-inflammatory/immune suppressant medication for >7 days within the past 30 days prior to entry
* pregnant or breastfeeding
* eGFR < 60 ml/min/1.73 m2 calculated by 2021 CKD-EPI Creatinine
* known severe allergy to iodinated contrast media (CCTA), dextrans/DTPA/radiometals (99mTc-tilmanocept SPECT/CT), or regadenoson/adenosine (cardiac PET/CT).
* self-reported significant radiation exposure (>2 CT angiograms) received within the past 12 months
* concurrent enrollment in conflicting research study.

Non-HIV-infected women:

As above, save for addition of inclusion criteria for negative HIV test and absent inclusion criteria for HIV and self-report of stable ART.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Women with HIV and women without HIV
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Coronary flow reserve on Cardiac PET | Baseline

SECONDARY OUTCOMES:
Arterial inflammation on 99mTc-tilmanocept SPECT/CT | Baseline
Atherosclerotic plaque on Contrast Enhanced Coronary and Aortic Computed Tomography Angiography | Baseline
Fractional Flow Reserve | Baseline
Markers of inflammation/immune activation | Baseline
Markers of endothelial dysfunction | Baseline
Markers of mitochondrial disease/dysfunction | Baseline
Markers of myocardial stretch/injury | Baseline
Hormonal/metabolic parameters | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Markella V. Zanni, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided